CLINICAL TRIAL: NCT05396131
Title: The Use of Aeriseal ® in the Management of Collateral Ventilation Positive COPD Patients Undergoing ELVR (Endoscopic Lung Volume Reduction) Utilizing Endobronchial Valves
Brief Title: The Use of Aeriseal ® in the Management of Collateral Ventilation Positive COPD Patients Undergoing ELVR Utilizing Endobronchial Valves.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-MCVP-COPD-ELVR
Record Dates: First submitted 2021-09-20; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants diagnosed as either Collateral Ventilation (CV) Negative or CV Positive.
  CV Negative participants will only receive the endobronchial valves (EBV). CV Positive participants will receive both the lung sealant and the EBV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Collateral Ventilation Negative (Active Comparator): Collateral Ventilation Negative participants will have endobronchial valve implant
  Interventions: Device: Endobronchial Valve (EBV)
- Collateral Ventilation Positive (Experimental): Collateral Ventilation Positive participants will have the lung sealant applied and the endobronchial valve implant
  Interventions: Device: Lung Sealant; Device: Endobronchial Valve (EBV)

INTERVENTIONS:
Device: Lung Sealant — The Aeriseal System uses a polymer foam to block or seal fissures, peripheral airways, alveoli, and collateral channels to achieve lung volume reduction.
  Other Names: AeriSeal
  Arms: Collateral Ventilation Positive
Device: Endobronchial Valve (EBV) — The Zephyr EBV System are one way valves inserted into the airways to reduce lung hyperinflation.
  Other Names: Zephyr Endobronchial Valve System

SUMMARY:
The aim of this study is to determine the feasibility of combining a lung sealant with endobronchial valves EBV in managing patients with COPD who are collateral ventilation (CV) positive. This study has two arms; arm 1 is for CV positive participants who will receive the lung sealant and EBV; arm 2 is the CV negative group who will only receive EBV as the standard management.

ELIGIBILITY:
Inclusion Criteria:

* i. 18-85 years of age
* ii. Forced Expiratory Volume in 1second (FEV1) 20 - 50%
* iii. Residual Volume (RV) > 175%
* iv. 6 min walk test > 150 m
* v. Completed a course of Pulmonary rehabilitation
* vi. STRATX assessment - Left Upper Lobe as the most appropriate lobe to target for ELVR
* vii. This study will be investigating heterogenous emphysema only. Minimum of 15% differential in emphysema destruction scores at -950 HU

Exclusion Criteria:

* i. Acute uncontrolled medical illness including ischemic heart disease, cardiac failure, acute renal impairment
* ii. Acute respiratory tract infections
* iii. Significant bronchiectasis,
* iv. Co-existing interstitial lung diseases, pneumothorax,
* v. Known active malignancy
* vi. Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants converted from Collateral Ventilation positive (CV+) to Collateral Ventilation negative (CV-) | 4 weeks post lung sealant application
  Collateral ventilation status will be functionally assessed and confirmed via CHARTIS® System. Examination of left upper lobe to determine percentage of participants converted from collateral ventilation positive to a collateral ventilation negative state

SECONDARY OUTCOMES:
Number of participants with improved lung functioning as measured by lung function tests | 12weeks and 52 weeks post valve implant
  Lung function will be assessed by spirometry, plethysmography, lung diffusion capacity and capillary blood test
Changes Lung volume | 12weeks and 52 weeks post valve implant
  Changes in lung volume will be assessed using high resolution computed tomography (HRCT) and target lobe volume reduction (TLVR)

CONTACTS AND LOCATIONS:
Overall Officials: Alvin J Ing, MBBS, MD, FRACP, Principal Investigator — Clinical Professor and Respiratory Physician
Locations (1):
- Macquarie University, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ing AJ, Jayapadman A, Kim WV, Ly C, Ho-Shon K, Lilburn P, Carew A, Ng BJH, Saghaie T, Williamson JP. Reversal of collateral ventilation using endoscopic polymer foam in COPD patients undergoing endoscopic lung volume reduction with endobronchial valves: A controlled parallel group trial. Respirology. 2022 Dec;27(12):1064-1072. doi: 10.1111/resp.14338. Epub 2022 Aug 2. PMID 35918295